

October 18, 2022

# To: ClinicalTrials.gov

This is a cover page to the redacted SAP for APC-003 titled Phase 2 Double-Blind Placebo-Controlled 4-Period Single-Dose Crossover Factorial Study to Evaluate the Contribution of the Individual Drug Components to the Efficacy of the Combination of Atomoxetine and Roxybutynin in Obstructive Sleep Apnea.

The APC-003 SAP is associated with NCT04580394.

The following proprietary information was redacted from the SAP for APC-003:

- IND number
- Reference to the CRO (Contract Research Organization).

# Sincerely,



# Jeanne Brittain

Director, Program Management

| Quality Approval: | | | |
|---|---|---|---|
| Name | Title | Signature | Date |
| Francesca | Senior Director, GXP | DocuSigned by: | 10/19/2022 |
| Kelvy | Quality Assurance | Francisca Edwy Signer Name: Francesca Kelvy Signing Reason: I approve this document Signing Time: 10/19/2022 8:30:24 AM ED 35E78DD6A7F34F8AA557BB15D08339E | |



Phase 2 Randomized Double-Blind Placebo-Controlled 4-Period Single-Dose Crossover Factorial Study to Evaluate the Contribution of the Individual Drug Components to the Efficacy of the Combination of Atomoxetine and R-oxybutynin in Obstructive Sleep Apnea

| Protocol Number: | APC-003 |
|-------------------|-----------------|
| Protocol Version: | 2.0 |
| Protocol Date: | 06 January 2021 |

STATISTICAL ANALYSIS PLAN

Version 2.0



Phase 2 Randomized Double-Blind Placebo-Controlled 4-Period Single-Dose Crossover Factorial Study to Evaluate the Contribution of the Individual Drug Components to the Efficacy of the Combination of Atomoxetine and R-oxybutynin in Obstructive Sleep Apnea

#### STATISTICAL ANALYSIS PLAN

Version 2.0



**Author:** 

7AB7AB9F099E4A60867CB1F0B820EACB Bryce Weaver Biostatistician, CTI

DocuSigned by:





Rachael Gilbert Runyan Manager, Biostatistics, CTI



# **Sponsor Approval:**

Ronald Farkas Chief Medical Officer Apnimed, Inc.

Note that the last signature date is the effective date of the plan.




# **Table of Contents**

| LI | ST OF ABBRE | EVIATIONS AND TERMS | . 5 |
|---|---|---|---|
| 1. | INTRODUC | ΓΙΟΝ | . 7 |
| 2. | OBJECTIVE | S AND ENDPOINTS | . 7 |
| 2 | 2.1. Objectiv | ES | . 7 |
| | | y Objective | |
| | • | ary Objectives | |
| | 2.1.3. Explore | atory Objective | . 7 |
| 2 | | ΓS | |
| | 2.2.1. Primar | y Endpoint | . 8 |
| | 2.2.2. Second | ary Endpoints | . 8 |
| | 2.2.3. Explore | atory Endpoints | . 8 |
| | 2.2.4. Safety I | Endpoints | . 9 |
| 3. | INVESTIGA | TIONAL PLAN | . 9 |
| 3 | 3.1. STUDY DI | ESIGN | . 9 |
| 3 | 3.2. Treatme | NT | 10 |
| | 3.2.1. Randon | nization Scheme and Treatment Arm Assignment | 10 |
| | | g | |
| | | Schedule | |
| | _ | reatment Compliance | |
| 4. | GENERAL C | CONSIDERATIONS FOR DATA ANALYSIS | 11 |
| 2 | <b>4.1. D</b> ата <b>Q</b> U | ALITY ASSURANCE | 11 |
| 4 | | S SETS | |
| | 4.2.1. Enrolle | ed Set | 12 |
| | 4.2.2. Modifie | ed Intent-To-Treat Analysis (mITT) Set | 12 |
| | 4.2.3. Safety S | Set | 12 |
| | 4.2.4. Per Pro | otocol (PP) Set | 12 |
| 2 | 4.3. Assessmi | ENT WINDOWS | 12 |
| 4 | 4.4. HANDLIN | G OF DROPOUTS OR MISSING DATA | 12 |
| | 4.4.1. PSG Pa | arameters | 12 |
| | 4.4.2. DSST S | Scores | 13 |
| 4 | 4.5. Multipli | E COMPARISONS | 13 |
| 4 | 4.6. DATA DE | RIVATIONS AND TRANSFORMATIONS | 13 |
| 4 | 4.7. Repeatei | D MEASURE MODELING FOR SELECT ENDPOINTS | 13 |
| 5. | STUDY PAR | TICIPANTS | 14 |
| 4 | 5.1. Dispositi | ON OF PARTICIPANTS | 14 |
| 4 | 5.2. Protoco | L DEVIATIONS | 14 |



| Demographic | 14 |
|---|---|
| BASELINE CHARACTERISTICS | 14 |
| MEDICAL HISTORY | 15 |
| PRIOR AND CONCOMITANT MEDICATIONS | 15 |
| FICACY ANALYSIS | 15 |
| PRIMARY AND SECONDARY EFFICACY ANALYSIS OF HB(4%) | 15 |
| ADDITIONAL SECONDARY EFFICACY ANALYSIS | 16 |
| P.1. AHI(4%) | 16 |
| P.2. ODI(4%) | 16 |
| $P.3.$ Total time with $SaO_2 < 90\%$ | 16 |
| ?.4. Proportion of participants with $\geq 50\%$ reduction | 16 |
| EXPLORATORY EFFICACY ANALYSES | 17 |
| FETY ANALYSIS | 17 |
| EXTENT OF EXPOSURE | 17 |
| ADVERSE EVENTS | 17 |
| 2.1. Treatment-emergent Adverse Events | 18 |
| 2.2. Adverse Event Intensity | 18 |
| 2.3. Adverse Event Relationship to Study Medication | 18 |
| 2.4. Serious Adverse Events | 19 |
| 2.5. Adverse Event Summaries | 19 |
| VITAL SIGNS | 20 |
| DSST | 20 |
| PSG Parameters | 20 |
| TERIM ANALYSIS | 20 |
| MPLE SIZE AND POWER CALCULATIONS | 20 |
| PPENDICES | 21 |
| APPENDIX A: SCHEDULE OF ACTIVITIES | 21 |
| APPENDIX B: PROTOCOL-REQUIRED SAFETY LABORATORY ASSESSMENTS | 22 |
| | PRIMARY AND SECONDARY EFFICACY ANALYSIS OF HB(4%) |



# LIST OF ABBREVIATIONS AND TERMS

**Abbreviation Definition** 

AHI apnea-hypopnea index

AE adverse event

ATC anatomical, therapeutic, and chemical

CI confidence interval

CRO contract research organization

CSR clinical study report

DSST digit symbol substitution test

ECG electrocardiogram

eCRF electronic case report form(s)

EDC electronic data capture

HB hypoxic burden

HR heart rate

ICF informed consent form

LS least square

MedDRA medical dictionary for regulatory activities

mITT modified intent to treat

NAW number of awakenings

NREM non-rapid eye movement

ODI oxygen desaturation index

OSA obstructive sleep apnea

PP per protocol

PSG polysomnography

PT preferred term

REM rapid eye movement




| <b>Abbreviation</b> | <b>Definition</b> |
|---------------------|----------------------------------|
| SAE | serious adverse event |
| SaO <sub>2</sub> | oxygen saturation |
| SAP | statistical analysis plan |
| SD | standard deviation |
| SE | sleep efficiency |
| SOC | system organ class |
| SOL | sleep onset latency |
| TEAE | treatment-emergent adverse event |
| TST | total sleen time |

TST total sleep time

WASO wake after sleep onset

WHO world health organization




#### 1. INTRODUCTION

This statistical analysis plan (SAP) is based on the Protocol # APC-003 Version 2.0, dated 06 January 2021, titled "Phase 2 Randomized Double-Blind Placebo-Controlled 4-Period Single-Dose Crossover Factorial Study to Evaluate the Contribution of the Individual Drug Components to the Efficacy of the Combination of Atomoxetine and R-oxybutynin in Obstructive Sleep Apnea." AD109 is a new fixed-dose combination of atomoxetine and R-oxybutynin being developed for obstructive sleep apnea (OSA). Study APC-003 is designed to compare the efficacy of AD109 to placebo and the individual components of AD109, atomoxetine and R-oxybutynin, in OSA.

This document details the statistical methods planned to perform the final analyses of this study.

#### 2. OBJECTIVES AND ENDPOINTS

# 2.1. Objectives

# 2.1.1. Primary Objective

The primary objective is to evaluate the efficacy of AD109 compared to placebo as measured by the 4% definition of hypoxic burden (HB).

# 2.1.2. Secondary Objectives

The secondary objectives include:

- To evaluate the efficacy of AD109 compared to R-oxybutynin alone as measured by HB(4%)
- To evaluate the efficacy of AD109 compared to atomoxetine alone as measured by HB(4%)
- To evaluate the efficacy of AD109 compared to the other 3 study treatments as measured by the 4% definition for hypopneas (AHI).
- To evaluate the efficacy of AD109 compared to the other 3 study treatments as measured by the 4% definition of oxygen desaturation index (ODI).
- To evaluate the efficacy of AD109 compared to the other 3 study treatments as measured by total time with  $SaO_2 < 90\%$ .
- To evaluate the efficacy of AD109 compared to the other 3 study treatments on the proportion of participants with  $\geq$ 50% reduction in AHI, HB and ODI.

# 2.1.3. Exploratory Objective

The exploratory objectives are to evaluate the effects of AD109 compared to the other 3 study treatments on:

- Snoring index
- Sleep stages distribution and percentage of time in the various sleep stages
- Arousal index
- Fraction of hypopneas




• Alternative measures of AHI, ODI and HB

An additional exploratory objective is to evaluate the effects of AD109 compared to the other study treatments in the subgroup of participants meeting "moderate collapsibility" polysomnography (PSG) criteria at baseline (PSG-0).

# 2.2. Endpoints

# 2.2.1. Primary Endpoint

The primary efficacy endpoint is as follows:

• Change in log<sub>10</sub>(HB[4%] + 1), (scored in reference to AHI[4%]), AD109 vs. placebo

# 2.2.2. Secondary Endpoints

The secondary efficacy endpoints are as follows:

- Change in  $log_{10}(HB[4\%] + 1)$ , AD109 vs. R-oxybutynin alone
- Change in  $log_{10}(HB[4\%] + 1)$ , AD109 vs. atomoxetine alone
- Change in AHI(4%), AD109 vs. other 3 study treatments
- Change in ODI(4%), AD109 vs. the other 3 study treatments
- Total time with SaO<sub>2</sub><90%, PSG nights
- Proportion of participants with  $\geq 50\%$  reduction, AHI(4%), HB(4%), and ODI(4%)

#### 2.2.3. Exploratory Endpoints

The exploratory efficacy endpoints are as follows:

- PSG sleep and arousal parameters
  - o Sleep stages distribution and percentage of time in the various sleep stages
    - Sleep Efficiency (SE)
    - Wake After Sleep Onset (WASO)
    - Number of Awakenings (NAW)
    - Sleep Onset Latency (SOL)
    - Percentage of total sleep time (TST) spent in sleep stage N1 (Stage N1%)
    - Percentage of TST spent in sleep stage N2 (Stage N2%)
    - Percentage of TST spent in sleep stage N3 (Stage N3%)
    - Percentage of TST spent in sleep stage R (Stage R%)
  - Snoring index
  - Arousal indices (respiratory and spontaneous)
  - Fraction of hypopneas




- Alternate measures of AHI, ODI and HB
  - o AHI(4%) in non-rapid eye movement (NREM) sleep
  - o AHI(4%) in rapid eye movement (REM) sleep
  - o AHI(4%) adjusted for position
  - o AHI(3% or arousal)
  - o HB(3% or arousal)
  - o HB(Total)
  - o ODI(3%)
- Subgroup analyses of efficacy endpoints in participants meeting "moderate collapsibility" criteria (AHI[4%] 10 to <20, or AHI[4%] ≥20 if any one of the following are met: F<sub>hypopnea</sub> of >90% OR mean oxygen desaturation of obstructive events of ≤4% OR F<sub>hypopnea</sub> of 50 to 90% and mean oxygen desaturation of 4 to 8%) at baseline (PSG-0).

# 2.2.4. Safety Endpoints

The safety endpoints are as follows:

- Physical exam, vital signs, clinical laboratory assessment
- Spontaneous adverse events, including the post-dosing period
- Digit Symbol Substitution Test (DSST)
- PSG parameters:
  - Total sleep time (TST)
  - Heart rate (HR)
  - o Total time with SaO<sub>2</sub><90%

## 3. INVESTIGATIONAL PLAN

# 3.1. Study Design

Study APC-003 is a double-blind, placebo-controlled, 4-period, single-dose crossover study designed to compare the efficacy of AD109 to placebo and the individual components of AD109 (atomoxetine and R-oxybutynin).

A total of 58 participants will be enrolled. Patients who meet all enrollment criteria will be randomized to receive the following experimental treatments, one treatment on each of 4 PSG nights:

- A: Atomoxetine 75 mg + R-oxybutynin 2.5 mg (AD109)
- B: Atomoxetine 75 mg
- C: R-oxybutynin 2.5 mg
- D: Placebo




Dosing of the study treatment will occur immediately prior to lights out. Each morning following PSG exams in the crossover period the DSST will be administered.

Each PSG night is followed by a 1-week washout period. Adverse event (AE) and serious adverse event (SAE) information is recorded at each study visit and by telephone contact with participants during each washout period and at the end of the final washout period. Overall study duration will be up to 10 weeks (see Figure 1).

Figure 1: Overview of Study Design



PSG = polysomnography

#### 3.2. Treatment

Study treatment is defined as any investigational treatment(s), marketed product(s), placebo, or medical device(s) intended to be administered to a study participant according to the study protocol.

Two capsules are taken each night of drug treatment, either:

- 1 capsule of atomoxetine 75 mg + 1 capsule of R-oxybutynin 2.5 mg
- 1 capsule of atomoxetine 75 mg and 1 capsule of placebo
- 1 capsule of R-oxybutynin 2.5 mg and 1 capsule of placebo
- 2 capsules of placebo

Study medication is taken immediately prior to lights out.

# 3.2.1. Randomization Scheme and Treatment Arm Assignment

The randomization scheme will allocate participants to one of the following 24 treatment sequences: ABCD, ABDC, ACBD, ACDB, ADBC, ADCB, BACD, BADC, BCAD, BCDA, BDAC, BDCA, CABD, CADB, CBAD, CBDA, CDAB, CDBA, DABC, DACB, DBAC, DBCA, DCAB, DCBA (using treatments A, B, C, and D as defined in Section 3.1).

Participants who withdraw from the study will not be replaced.




### 3.2.2. Blinding

The investigator, study personnel and participant will be blinded to the identity of the study drug in all treatment periods. The CRO staff dealing with blinded site study staff will also be blinded. The Sponsor, Medical Monitor, CRO's Drug Safety and Pharmacovigilance staff, as well as site personnel required for drug administration will also be blinded. The centralized PSG technologists will be blinded to treatment assignment.

The CTI unblinded statistician who reviews the production randomization list will be unblinded to the treatment sequence a participant receives; however, this individual will not have access to study data prior to study completion. The investigational pharmacist and/or the study coordinator, depending on the site, will be unblinded to treatment assignment for the purposes of preparing, controlling, dispensing study product and documenting accountability of study product.

# 3.2.3. Dosing Schedule

There are 4 randomized crossover PSG nights. Each PSG night is followed by a 1-week washout period. Dosing of the study treatment will occur immediately prior to lights out.

# 3.2.4. Study Treatment Compliance

Only participants enrolled in the study treatments and only authorized site staff may supply or administer study treatments.

After receiving Sponsor approval in writing, sites are responsible for returning all unused or partially used study treatment to the Sponsor or designated third party or for preparing the study treatment for destruction vis incineration. Unused study drug will be counted and recorded by study personnel to assess study treatment compliance.

#### 4. GENERAL CONSIDERATIONS FOR DATA ANALYSIS

In general, continuous variables will be summarized by presenting the sample size (N), number of participants with available data (n), mean, standard deviation (SD), median, minimum, and maximum. In summaries of change from baseline safety variables, only participants with both baseline and post baseline data will be included. Categorical variables will be summarized by presenting the number and percentage of participants within each category. Calculation of percentages will exclude missing data as a category. Where appropriate, descriptive statistics may be presented with 95% confidence intervals (CIs).

All tabulations will be based on pooled data across centers.

The data analyses will be performed using SAS for Windows, version 9.4 or higher (SAS, Cary, NC), except where other software may be deemed more appropriate.

CTI Clinical Trial and Consulting Services (Covington, KY) will perform the efficacy and safety analyses. Apnimed, Inc., will perform subgroup analyses of efficacy endpoints in participants meeting "moderate collapsibility" criteria described in Section 2.2.3. Any changes to the analyses that are not included in this SAP will be documented in the clinical study report (CSR).

#### 4.1. Data Quality Assurance

Once all the source verification is complete, all queries are resolved, and the database has been




updated appropriately, the database will be locked and made available to CTI Biostatistics for final analysis.

Data may be made available to CTI Biostatistics for programming purposes prior to database lock at a time when source verification and query resolution is ongoing.

All SAS programs used to create analysis data sets, tables, and listings will be independently programmed by two individuals. The independent SAS outputs produced will be compared, and the SAS programs will be updated until the outputs match.

# 4.2. Analysis Sets

#### 4.2.1. Enrolled Set

The Enrolled Set is defined as all participants who signed the informed consent form (ICF) (including screening failures).

# 4.2.2. Modified Intent-To-Treat Analysis (mITT) Set

The mITT Set comprises all participants who are randomized, take at least 1 dose of any of the study treatments, and have at least 1 measurement on the primary endpoint.

Participants will be analyzed for efficacy according to the randomly assigned treatment for each period.

# 4.2.3. Safety Set

The Safety Set consists of all participants who are randomized and receive at least 1 dose of any of the study treatments. Participants will be analyzed for safety based on the treatment received for each period. Treatment received is defined as the actual treatment taken during each period.

### 4.2.4. Per Protocol (PP) Set

The PP Set consists of all participants without any major protocol violations that could influence efficacy assessment. Participants in this set will be analyzed according to the treatment they received for each period. Treatment received is defined as the actual treatment taken during each period.

# 4.3. Assessment Windows

Data will be summarized by the eCRF (Study Visit) in which it was collected as long as the data is within the windows specified.

# 4.4. Handling of Dropouts or Missing Data

Missing data will remain missing. No imputation of missing data will be performed.

# 4.4.1. PSG Parameters

The criteria for use of PSG data will be as follows:

• When TST is < 120 minutes, only TST, time in bed, Stage N1%, Stage N2%, Stage N3%, and Stage R% will be reported. All other PSG indices will be excluded.




- Any AHI and HB parameters during REM will be reported only when the time spent in REM is > 5 minutes.
- Any AHI and ODI parameters in supine position will be reported only when the time spent supine is > 5 minutes.

#### 4.4.2. DSST Scores

A DSST total correct of 0 will be dropped from the repeated measures model.

# 4.5. Multiple Comparisons

Each group of endpoints for this study contains three hypothesis tests based on the study treatment: i) AD109 vs placebo, ii) AD109 vs R-oxybutynin, iii) AD109 vs atomoxetine. The type I error will be controlled by a fixed sequence procedure in which the hypothesis tests are conducted in the following order: i) AD109 vs placebo, ii) AD109 vs R-oxybutynin, iii) AD109 vs atomoxetine. Primary and secondary endpoints will be tested sequentially in the order they appear in Section 2.2.1 and Section 2.2.2. All hypothesis tests will test that the two-sided p-value is less than 0.05. All hypothesis tests for secondary endpoints will also be reported using the nominal 0.05 two-sided alpha level.

#### 4.6. Data Derivations and Transformations

Study Day will be calculated as:

- Date of assessment date of randomization + 1 for assessments done on or after date of randomization
- Date of assessment date of randomization for assessments done before date of randomization

For each efficacy and safety endpoint, the baseline value will be calculated as the last non-missing value prior to randomization (except where unscheduled assessments are performed the baseline value should be the value recorded at Screening). Where applicable, change from baseline values will be calculated as:

Change from Baseline = assesment value – baseline value,

while the percent change from baseline values will be calculated as:

percent change from baseline = 
$$\frac{\text{change from baseline}}{\text{baseline value}} \times 100\%$$
.

For the endpoints that look for the proportion of participants with  $\geq 50\%$  reduction, participants will be assigned a visit level indicator:

Indicator of 
$$\geq 50\%$$
 reduction = 
$$\begin{cases} 1 & \text{if percent change from baseline } \leq -50\% \\ 0 & \text{otherwise} \end{cases}$$

# 4.7. Repeated Measure Modeling for Select Endpoints

In Section 6, modeling will be used for comparisons between study treatments with respect to given endpoints using the PROC GLIMMIX procedure in SAS. The model will include study treatment and visit as fixed effects. Within participant variability (nested within treatment




sequence) will be modeled using an unstructured (e.g., TYPE = UN, CHOL) covariance pattern. The unstructured covariance parametrized through its Cholesky root is to be used for logistic regression models and models in which convergence fails for the completely unstructured covariance. Point estimates (e.g., mean, difference of means) and inferential statistics (e.g., confidence interval, p-values) will provided be estimated using least square (LS) methods. Unless otherwise stated, the link will be identity and the distribution gaussian.

#### 5. STUDY PARTICIPANTS

# 5.1. Disposition of Participants

A table of frequency counts and percentages of all participants who are enrolled, randomized, and included in each analysis set will be provided. Participant disposition including study completion status and reasons for early termination will be tabulated overall. A by-participant listing will be provided.

#### **5.2.** Protocol Deviations

Two separate by-participant listings for major and minor protocol deviations will be provided.

### 5.3. Demographic

Descriptive statistics will be used to summarize the demographic characteristics (age, gender, race, ethnicity, height, weight, and BMI) overall using the Safety Set. A by-participant listing will also be provided.

#### **5.4.** Baseline Characteristics

The results of the following assessments completed during the baseline PSG (PSG-0) will be summarized overall using the Safety Set:

- AHI(4%)
- ODI(4%)
- HB(4%)
- Total time with SaO<sub>2</sub> < 90%
- Snoring index
- Arousal indices (respiratory and spontaneous)
- Fraction of hypopneas
- WASO
- Sleep stage (N1, N2, N3, R) separately in minutes and percent of total sleep time
- Sleep efficiency
- Number of awakenings
- Sleep onset latency




- Heart rate
- Total sleep time
- Systolic blood pressure
- Diastolic blood pressure

Additionally, the Epworth sleepiness scale total score will be summarized.

A by-participant listing will also be provided for Epworth sleepiness scale. The baseline PSG parameters and vital signs will be included in their respective general listings.

# 5.5. Medical History

All medical conditions and surgical procedures will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) version 23.0. The number and percent of participants with each medical condition and surgical procedure will be presented by MedDRA system organ class (SOC), preferred term (PT) overall for the Safety Set. Each participant will be counted only once per SOC and PT. A by-participant listing will also be provided.

#### 5.6. Prior and Concomitant Medications

Prior and concomitant medications will be coded using the September 2020 B3 Global World Health Organization (WHO) Drug Dictionary version. The number and percent of participants using each medication will be tabulated by Anatomical Therapeutic Chemical (ATC) level 3 and preferred name overall. Each prior or concomitant medication reported more than one time will only be counted once per participant for each ATC level and preferred name. A by-participant listing will also be provided.

#### 6. EFFICACY ANALYSIS

The mITT Set will be used for all efficacy analyses.

# 6.1. Primary and Secondary Efficacy Analysis of HB(4%)

Comparisons will be performed as described in Section 4.5. A repeated measures model (see Section 4.7) will be used to model change in  $\log_{10}(HB[4\%] + 1)$  from baseline. Model based LS mean estimates will be provided for the following:

- mean change from baseline by study treatment (AD109, placebo, R-oxybutynin, and atomoxetine),
- difference in mean change between AD109 and the other three treatments (placebo, Roxybutynin, and atomoxetine) with 95% confidence interval and respective p-values (for the null hypothesis).

If the model shows there is a visit (i.e., period) effect, then ad hoc analyses will be performed. A sensitivity analysis will be performed using the PP Set on the primary efficacy endpoint using the same methods described above and using HB(4%) with identity transform (i.e., without transform) on the mITT set.

Descriptive statistics for the reported log<sub>10</sub>(HB[4%] + 1) value and change from baseline in




 $log_{10}(HB[4\%] + 1)$  will be presented by study treatment. By taking the inverse transformations of the respective means, the geometric mean of HB(4%) + 1 and the ratio of the geometric mean to baseline will be reported.

# 6.2. Additional Secondary Efficacy Analysis

# 6.2.1. **AHI(4%)**

Multiple comparisons will be performed as described in Section 4.5. A repeated measures model will be used to model change in AHI(4%) from baseline. Model based LS mean estimates will be provided for the following:

- mean change by study treatment (AD109, placebo, R-oxybutynin, and atomoxetine),
- difference in mean change between AD109 and the other three treatments (placebo, Roxybutynin, and atomoxetine) with 95% confidence interval and respective p-values (for the null hypothesis).

Descriptive statistics for the reported AHI(4%) value and change from baseline in AHI(4%) will be presented by study treatment.

# 6.2.2. **ODI**(4%)

Multiple comparisons will be performed as described in Section 4.5. A repeated measures model will be used to model change in ODI(4%) from baseline. Model based LS mean estimates will be provided for the following:

- mean change by study treatment (AD109, placebo, R-oxybutynin, and atomoxetine),
- difference in mean change between AD109 and the other three treatments (placebo, Roxybutynin, and atomoxetine) with 95% confidence interval and respective p-values (for the null hypothesis).

Descriptive statistics for the reported ODI(4%) value and change from baseline in ODI(4%) will be presented by study treatment.

#### 6.2.3. Total time with SaO<sub>2</sub><90%

Multiple comparisons will be performed as described in Section 4.5. A repeated measures model will be used to model change in total time with SaO2<90% from baseline. Model based LS mean estimates will be provided for the following:

- mean change by study treatment (AD109, placebo, R-oxybutynin, and atomoxetine),
- difference in mean change between AD109 and the other three treatments (placebo, R-oxybutynin, and atomoxetine) with 95% confidence interval and respective p-values (for the null hypothesis).

Descriptive statistics for the reported total time with SaO<sub>2</sub><90% value and change from baseline in total time with SaO<sub>2</sub><90% will be presented by study treatment.

# 6.2.4. Proportion of participants with ≥50% reduction

Three separate repeated measures models (see section 4.7) will be used to model the probability




of a  $\geq$ 50% reduction in HB(4%), AHI(4%), and ODI(4%) values respectively. A logit link with binomial distribution will be employed. For each of the three endpoints, model based LS mean estimates will be provided for the following:

• odds ratios for a ≥50% reduction for AD109 vs the other three treatments (placebo, Roxybutynin, and atomoxetine) with 95% confidence intervals and respective p-values (for null hypothesis).

The proportion, with 95% CI, of participants with  $\geq$ 50% reduction in HB(4%), AHI(4%), and ODI(4%) will be presented by study treatment in the same table as the models.

# **6.3.** Exploratory Efficacy Analyses

Descriptive statistics for the reported value and change from baseline by study treatment will be reported for sleep stages distribution and percentage of time in the various sleep stages (SE, WASO, NAW, SOL, Stage N1%, Stage N2%, Stage N3%, Stage R%). A 95% confidence interval will be included for the change from baseline.

Snoring index, arousal indices (respiratory and spontaneous), fraction of hypopneas (see below) and alternate measures of AHI, ODI, and HB (AHI[4%]: in NREM sleep, in REM sleep, AHI adjusted for position [see below]; AHI[3% or arousal]; HB[3% or arousal]; HB[Total]; ODI[3%]) and will have results provided similar to Section 6.1 (including the model of change from baseline and the descriptive statistics).

Additional clarifying details for the analysis of some of these endpoints is as follows:

- Fraction of hypopneas will be calculated by using the number of hypopneas divided by the total number of apneas plus hypopneas.
- AHI adjusted for position: An additional covariate of % time supine (%TS) will be added to the repeated measures model for AHI(4%).

#### 7. SAFETY ANALYSIS

Safety assessments will include measurement of adverse events (AEs) and serious AEs (SAEs).

The analyses will be descriptive and will be based on the Safety Set. The safety assessments will be summarized by the treatment the participant actually received within each period.

# 7.1. Extent of Exposure

The number and percentage of participants receiving study treatment will be summarized by study treatment and overall. A by-patient listing will be provided.

#### 7.2. Adverse Events

An AE is any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the medicinal product.

An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study treatment.




# 7.2.1. Treatment-emergent Adverse Events

A treatment-emergent adverse event (TEAE) is defined as any event not present prior to exposure of study drug or an event already present that worsens in either severity or frequency following exposure. Each TEAE is assigned to the most recent study treatment administered on or before the TEAE's date of onset.

# 7.2.2. Adverse Event Intensity

The Investigator will make an assessment of intensity for each AE and SAE reported during the study and assign it to one of the following categories:

- Mild: An event that is easily tolerated by the participant, causing minimal discomfort and not interfering with everyday activities.
- Moderate: An event that causes sufficient discomfort and interferes with normal everyday activities.
- Severe: An event that prevents normal everyday activities. An AE that is assessed as severe should not be confused with an SAE. Severe is a category utilized for rating the intensity of an event; and both AE and SAE can be assessed as severe.

An event is defined as 'serious' when it meets at least one of the predefined outcomes as described in the definition of an SAE, NOT when it is rated as severe.

# 7.2.3. Adverse Event Relationship to Study Medication

The Investigator is obligated to assess the relationship between study treatment and each occurrence of each AE/SAE.

- A "reasonable possibility" of a relationship conveys that there are facts, evidence, and/or arguments to suggest a causal relationship, rather than a relationship cannot be ruled out.
- The Investigator will use clinical judgment to determine the relationship.
- Alternative causes, such as underlying disease(s), concomitant therapy, and other risk factors, as well as the temporal relationship of the event to study treatment administration will be considered and investigated.
- The Investigator will also consult the Investigator's Brochure and/or Product Information, for marketed products, in his/her assessment.
- For each AE/SAE, the Investigator must document in the medical notes that he/she has reviewed the AE/SAE and has provided an assessment of causality.
- There may be situations in which an SAE has occurred and the Investigator has minimal information to include in the initial report to the CRO. However, it is very important that the Investigator always make an assessment of causality for every event before the initial transmission of the SAE data to the CRO.
- The Investigator may change his/her opinion of causality in light of follow-up information and send an SAE follow-up report with the updated causality assessment.
- The causality assessment is one of the criteria used when determining regulatory reporting requirements.




#### 7.2.4. Serious Adverse Events

An SAE is defined as any untoward medical occurrence that, at any dose:

- Results in death;
- Is life-threatening;
- Requires inpatient hospitalization or prolongation of existing hospitalization;
- Results in persistent disability/incapacity;
- Is a congenital anomaly/birth defect;
- Other situations.

#### 7.2.5. Adverse Event Summaries

Adverse event data will be displayed in listings by participant. The number and percentage of participants with AEs will be tabulated by SOC and PT. A participant with multiple AEs within a SOC or PT will be counted once toward the total for the total for the SOC or PT.

All AEs (serious and non-serious) occurring after completion of the informed consent process and before the end of study, regardless of relationship to study drug, will be included and presented by MedDRA SOC and PT.

For TEAEs, the following will be summarized by study treatment and presented for the Safety Set.

- i. An overall summary of TEAEs, which includes:
  - a. the number and percentage of participants experiencing any TEAE
  - b. the number and percentage of participants experiencing any TEAE by strongest relationship to study medication
  - c. the number and percentage of participants experiencing any TEAE by greatest intensity
  - d. the number and percentage of participants experiencing any TESAE
- ii. the number and percentage of participants experiencing any TEAE by SOC, PT
- iii. the number and percentage of participants experiencing any TEAE by SOC, PT and the greatest intensity
- iv. the number and percentage of participants experiencing any TEAE by SOC, PT and the strongest relationship to study medication
- v. the number and percentage of participants experiencing any TEAE leading to study discontinuation by SOC and PT.

In the overall summary of AEs table, besides tabulating the number and percentage of participants, the total number of AE episodes will also be provided. If a participant has repeated episodes of a particular AE within a treatment period, all episodes will be counted in the summary table and displayed by treatment.

For displays by SOC and PT, each participant will be counted only once per SOC and PT within each treatment.




All occurrences of all AEs will be listed for each participant, grouped by treatment. The listing will contain the following information: treatment sequence, treatment, verbatim term, SOC, PT, intensity, relationship to study medication, date and day of onset, date and day of resolution, treatment given to treat the adverse event, action taken, the outcome, whether the event was an SAE, whether it led to withdrawal. Listings will be sorted by treatment sequence, participant identification number, onset date, SOC, and PT. If onset year is non-missing but month and/or date is missing, then the day of the most recent study drug dose will be imputed as onset date.

# 7.3. Vital Signs

Vital sign data will be summarized by presenting descriptive statistics of actual values and changes from baseline by study treatment. Vital sign parameters include respiratory rate, temperature, systolic blood pressure, diastolic blood pressure, and heart rate. A by-participant listing of vital signs will also be provided.

#### **7.4. DSST**

A repeated measures model (see Section 4.7) will be used to model the natural log of total number of the correct symbol assignments<sup>1</sup> (log (total completed - total incorrect)) from the DSST.

Exponentiation of the model-based LS mean estimates of log values will be used to provide the following:

- Geometric mean of DSST by study treatment (AD109, placebo, R-oxybutynin, and atomoxetine), and
- Ratio of (geometric) mean of DSST between AD109 and the other three treatments (placebo, R-oxybutynin, and atomoxetine) with the 95% confidence intervals.

Descriptive statistics of DSST and a by-participant listing (with both raw values and natural log of total complete) will also be provided.

#### 7.5. PSG Parameters

PSG safety data will be summarized by presenting descriptive statistics of actual values and changes from baseline by treatment. PSG safety parameters include total sleep time, heart rate, and total time with SaO<sub>2</sub><90%. A by-participant listing of PSG parameters (including baseline and efficacy parameters) will also be provided.

#### 8. INTERIM ANALYSIS

No formal interim analysis is planned.

# 9. SAMPLE SIZE AND POWER CALCULATIONS

A total of 58 patients will enter the 4-treatment crossover study. The study will have 80% power to detect a treatment difference at a two-sided 0.05 significance level, if the true difference between treatments on HB is at least -3.7 %min/h. This assumes that the within-participant


<sup>&</sup>lt;sup>1</sup> In the case that the total correct is 0, the participant will be dropped from the model.



standard deviation is 9, estimated from Study APN-006, and that the discontinuation rate is less than 20%.

#### 10. **APPENDICES**

# 10.1. Appendix A: Schedule of Activities

| | Screeni | ng | | 4 | -Way C | rossovei | Perio | l Visit 3 | -6 | | End of Study Evaluation <sup>1</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedures | Daytime<br>V1 | PSG<br>V2 | PSG<br>V3 | Wash-<br>out <sup>2</sup> | PSG<br>V4 | Wash-<br>out | PSG<br>V5 | Wash-<br>out | PSG<br>V6 | Wash-<br>out | |
| Trial Day (Visit Window) | Up to 4 w | eeks | | | | Up to 8 | weeks | | | • | 2 weeks post V6 ± 3 days |
| Informed consent | X | | | | | | | | | | |
| Non-PSG enrollment criteria | X | | | | | | | | | | |
| Demography | X | | | | | | | | | | |
| ESS | X | | | | | | | | | | |
| Physical exam | X | | | | | | | | | | |
| Medical history | X | | | | | | | | | | |
| Clinical laboratory test | X | | | | | | | | | | |
| Pregnancy test <sup>3</sup> | X | | | | | | | | | | |
| 12 Lead ECG | X | | | | | | | | | | |
| PSG Exam | | X <sup>4</sup> | X | | X | | X | | X | | |
| Randomization <sup>5</sup> | | | X | | | | | | | | |
| Administration of study treatment <sup>6</sup> | | | X | | X | | X | | X | | |
| DSST <sup>7</sup> | | | X | | X | | X | | X | | |
| Vital signs <sup>8</sup> | X | X | X | | X | | X | | X | | |
| AE/SAE monitoring | | | X | X | X | X | X | X | X | X | X |
| Prior/concomitant medication monitoring | X | X | X | X | X | X | X | X | X | X | X |

Abbreviations: AE = adverse event; DSST = Digit Symbol Substitution Test; ECG = electrocardiogram; ESS = Epworth Sleepiness Scale; PSG = polysomnography; SAE = serious adverse event; WOCBP = women of childbearing potential.

 **CONFIDENTIAL** 

<sup>&</sup>lt;sup>1</sup> Can be conducted remotely. For patients enrolling in Study APC-003-OLE, can be conducted concurrently with first visit of Study APC-003-OLE. <sup>2</sup> Each washout period is a minimum of 7 days

<sup>3</sup> WOCBP only

<sup>&</sup>lt;sup>5</sup> Randomization occurs when participant meets enrollment criteria up to the time of the first crossover period

<sup>&</sup>lt;sup>6</sup> Study medication administered immediately before lights out

<sup>&</sup>lt;sup>7</sup> Administer at similar time after awakening after each crossover PSG, approximately 1 hour after awakening

<sup>&</sup>lt;sup>8</sup> Vital signs include the following: seated blood pressure, pulse, respiratory rate; vital signs on PSG nights taken after admission to PSG lab



# 10.2. Appendix B: Protocol-Required Safety Laboratory Assessments

| Laboratory<br>Assessments | Parameters | | |
|---|---|---|---|
| Hematology | Hematocrit<br>Hemoglobin<br>Platelet Count<br>RBC Count | RBC Indices (MCV,<br>MCH, MCHC) | WBC count with Differential |
| Serum Chemistry | Albumin BUN Creatinine Potassium Sodium Bilirubin Total Protein Uric acid | ALT AST Alkaline phosphatase Calcium Glucose Total cholesterol Chloride Bicarbonate | |
| Routine<br>Urinalysis | Specific gravity, bilirubin, color, appearance, leukocyte esterase, nitrite, pH, protein (albumin), glucose, ketones, occult blood, urobilinogen Microscopic examination (if positive protein, leukocyte esterase, blood or nitrite) | | |
| Other Tests | performed if need • Urine test of drug | nancy test at screening. | |

Abbreviations: ALT = alanine aminotransferase; AST = aspartate aminotransferase; BUN = blood urea nitrogen; HbA1c = hemoglobin A1c (glycated hemoglobin); hCG = human chorionic gonadotropin; RBC = red blood cell count; WBC= white blood cell; WOCBP = women of childbearing potential.


# **DocuSign**

#### **Certificate Of Completion**

Envelope Id: F85C8F878A2B4CCA9AB289D2ADF78005

Subject: Please DocuSign: APC-003 SAP v2.0.docx

Source Envelope:

Document Pages: 22 Signatures: 3
Certificate Pages: 5 Initials: 0

AutoNav: Enabled

**Envelopeld Stamping: Disabled** 

Time Zone: (UTC-05:00) Eastern Time (US & Canada)

Status: Completed

Envelope Originator: Bryce Weaver

100 E. RiverCenter Blvd

**Suite 1600** 

Covington, KY 41011 bweaver@ctifacts.com IP Address: 72.49.30.54

#### **Record Tracking**

Status: Original

5/13/2021 12:25:23 PM

Holder: Bryce Weaver

bweaver@ctifacts.com

Timestamp

Location: DocuSign

Sent: 5/13/2021 12:31:20 PM

Viewed: 5/13/2021 12:31:56 PM

Signed: 5/13/2021 12:34:27 PM

# **Signer Events**

Bryce Weaver bweaver@ctifacts.com

Biostatistician II

CTI Clinical Trial and Consulting Services- Part 11

Security Level: Email, Account Authentication

(Required)

#### Signature

Bryce Weaver

•

Signature Adoption: Pre-selected Style

Signature ID:

7AB7AB9F-099E-4A60-867C-B1F0B820EACB

Using IP Address: 72.49.30.54

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):

I am the author of this document

#### **Electronic Record and Signature Disclosure:**

Not Offered via DocuSign

Rachael Gilbert Runyan rrunyan@ctifacts.com Manager, Biostatistics

CTI Clinical Trial and Consulting Services Security Level: Email, Account Authentication

(Required)

Rachael Gilbert Runyan

Sent: 5/13/2021 12:31:20 PM Viewed: 5/13/2021 1:09:39 PM

Viewed: 5/13/2021 1:09:39 PM Signed: 5/13/2021 1:10:01 PM

Signature Adoption: Pre-selected Style

Signature ID:

5953F54F-F52D-42E0-9BA1-7E8D870EEDAB

Using IP Address: 74.215.68.242

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):

I approve this document

# Electronic Record and Signature Disclosure:

Not Offered via DocuSign

| Signer Events | Signature | Timestamp |
|---|---|---|
| Ronald Farkas | | Sent: 5/13/2021 12:31:20 PM |
| rfarkas@apnimed.com | Ronald Farkas | Viewed: 5/13/2021 12:47:45 PM |
| Chief Medical Officer | | Signed: 5/13/2021 12:51:13 PM |
| Ron Farkas | Signature Adoption: Pre-selected Style | |
| Security Level: Email, Account Authentication (Required) | Signature Adoption: Pre-selected Style | |
| | 2A5F46E3-93FC-40C7-8A20-AB4EF320DAB7 | |
| | Using IP Address: 71.179.160.191 | |
| | With Signing Authentication via DocuSign password | 1 |
| | With Signing Reasons (on each tab): | |
| | I approve this document | |

# Electronic Record and Signature Disclosure: Accepted: 7/17/2020 9:40:08 AM ID: 7410fab0-c816-4828-a4ed-9fb902e0e97a

| In Person Signer Events | Signature | Timestamp |
|---|---|---|
| Editor Delivery Events | Status | Timestamp |
| Agent Delivery Events | Status | Timestamp |
| Intermediary Delivery Events | Status | Timestamp |
| Certified Delivery Events | Status | Timestamp |
| Carbon Copy Events | Status | Timestamp |
| Witness Events | Signature | Timestamp |
| Notary Events | Signature | Timestama |
| <b>,</b> | Signature | Timestamp |
| Envelope Summary Events | Status | Timestamps |
| | - | · |
| Envelope Summary Events Envelope Sent Certified Delivered Signing Complete | Status Hashed/Encrypted Security Checked Security Checked | Timestamps 5/13/2021 12:31:20 PM 5/13/2021 12:47:45 PM 5/13/2021 12:51:13 PM |

#### ELECTRONIC RECORD AND SIGNATURE DISCLOSURE

From time to time, CTI Clinical Trial and Consulting Services (we, us or Company) may be required by law to provide to you certain written notices or disclosures. Described below are the terms and conditions for providing to you such notices and disclosures electronically through the DocuSign system. Please read the information below carefully and thoroughly, and if you can access this information electronically to your satisfaction and agree to this Electronic Record and Signature Disclosure (ERSD), please confirm your agreement by selecting the check-box next to 'I agree to use electronic records and signatures' before clicking 'CONTINUE' within the DocuSign system.

# **Electronic Signature Responsiblities**

You agree that your electronic signature is the equivalent of a hand-written signature and that you are responsible for actions initiated using your electronic signature. You agree to report unauthorized usage to CTI upon discovery of such usage via email to esign@ctifacts.com.

# Getting paper copies

At any time, you may request from us a paper copy of any record provided or made available electronically to you by us. You will have the ability to download and print documents we send to you through the DocuSign system during and immediately after the signing session and, if you elect to create a DocuSign account, you may access the documents for a limited period of time (usually 30 days) after such documents are first sent to you. After such time, if you wish for us to send you paper copies of any such documents from our office to you, you will be charged a perpage fee. You may request delivery of such paper copies from us by following the procedure described below.

# Withdrawing your consent

If you decide to receive notices and disclosures from us electronically, you may at any time change your mind and tell us that thereafter you want to receive required notices and disclosures only in paper format. How you must inform us of your decision to receive future notices and disclosure in paper format and withdraw your consent to receive notices and disclosures electronically is described below.

#### Consequences of changing your mind

If you elect to receive required notices and disclosures only in paper format, it will slow the speed at which we can complete certain steps in transactions with you and delivering services to you because we will need first to send the required notices or disclosures to you in paper format, and then wait until we receive back from you your acknowledgment of your receipt of such paper notices or disclosures. Further, you will no longer be able to use the DocuSign system to

receive required notices and consents electronically from us or to sign electronically documents from us.

# All notices and disclosures will be sent to you electronically

Unless you tell us otherwise in accordance with the procedures described herein, we will provide electronically to you through the DocuSign system all required notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to you during the course of our relationship with you. To reduce the chance of you inadvertently not receiving any notice or disclosure, we prefer to provide all of the required notices and disclosures to you by the same method and to the same address that you have given us. Thus, you can receive all the disclosures and notices electronically or in paper format through the paper mail delivery system. If you do not agree with this process, please let us know as described below. Please also see the paragraph immediately above that describes the consequences of your electing not to receive delivery of the notices and disclosures electronically from us.

# **How to contact CTI Clinical Trial and Consulting Services:**

You may contact us to let us know of your changes as to how we may contact you electronically, to request paper copies of certain information from us, and to withdraw your prior consent to receive notices and disclosures electronically as follows:

Please send an email to esign@ctifacts.com

# To advise CTI Clinical Trial and Consulting Services of your new email address

To let us know of a change in your email address where we should send notices and disclosures electronically to you, you must send an email message to us at esign@ctifacts.com and in the body of such request you must state: your previous email address, your new email address.

If you created a DocuSign account, you may update it with your new email address through your account preferences.

# To request paper copies from CTI Clinical Trial and Consulting Services

To request delivery from us of paper copies of the notices and disclosures previously provided by us to you electronically, you must send us an email to esign@ctifacts.com and in the body of such request you must state your email address, full name, mailing address, and telephone number.

# To withdraw your consent with CTI Clinical Trial and Consulting Services

To inform us that you no longer wish to receive future notices and disclosures in electronic format you may:

i. decline to sign a document from within your signing session, and on the subsequent page, select the check-box indicating you wish to withdraw your consent, or you may;

ii. send us an email to esign@ctifacts.com and in the body of such request you must state your email, full name, mailing address, and telephone number.

# Required hardware and software

The minimum system requirements for using the DocuSign system may change over time. The current system requirements are found here: <a href="https://support.docusign.com/guides/signer-guide-signing-system-requirements">https://support.docusign.com/guides/signer-guide-signing-system-requirements</a>.

# Acknowledging your access and consent to receive and sign documents electronically

To confirm to us that you can access this information electronically, which will be similar to other electronic notices and disclosures that we will provide to you, please confirm that you have read this ERSD, and (i) that you are able to print on paper or electronically save this ERSD for your future reference and access; or (ii) that you are able to email this ERSD to an email address where you will be able to print on paper or save it for your future reference and access. Further, if you consent to receiving notices and disclosures exclusively in electronic format as described herein, then select the check-box next to 'I agree to use electronic records and signatures' before clicking 'CONTINUE' within the DocuSign system.

By selecting the check-box next to 'I agree to use electronic records and signatures', you confirm that:

- You can access and read this Electronic Record and Signature Disclosure; and
- You can print on paper this Electronic Record and Signature Disclosure, or save or send this Electronic Record and Disclosure to a location where you can print it, for future reference and access; and
- Until or unless you notify CTI Clinical Trial and Consulting Services as described above, you consent to receive exclusively through electronic means all notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to you by CTI Clinical Trial and Consulting Services during the course of your relationship with CTI Clinical Trial and Consulting Services.